CLINICAL TRIAL: NCT04811092
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate Sotatercept When Added to Background Pulmonary Arterial Hypertension (PAH) Therapy in Newly Diagnosed Intermediate- and High-risk PAH Patients
Brief Title: Study of Sotatercept in Newly Diagnosed Intermediate- and High-Risk PAH Participants (MK-7962-005/A011-13)
Acronym: HYPERION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7962-005; A011-13 (Other: Acceleronpharma); MK-7962-005 (Other: MSD); 2023-509139-16 (Registry Identifier: EU CT); U1111-1309-6312 (Registry Identifier: UTN); 2021-000199-12 (EudraCT Number)
Record Dates: First submitted 2021-03-16; First posted 2021-03-23 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary; Hypertension; Sotatercept
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension | interventions — ACE-011

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo plus background PAH therapy (Placebo Comparator): Administered subcutaneously (SC) every 21 days plus background PAH therapy
  Interventions: Other: Placebo
- Sotatercept plus background PAH therapy (Experimental): Administered at a starting dose of 0.3 mg/kg, with a target dose of 0.7 mg/kg, subcutaneously (SC) every 21 days plus background PAH therapy
  Interventions: Drug: Sotatercept

INTERVENTIONS:
Drug: Sotatercept — Sotatercept (ACE-011) is a recombinant fusion protein consisting of the extracellular domain of the human activin receptor type IIA linked to the Fc piece of human IgG1
  Other Names: MK-7962; ACE-011
  Arms: Sotatercept plus background PAH therapy
Other: Placebo — Placebo
  Arms: Placebo plus background PAH therapy

SUMMARY:
The objective of this study is to evaluate the effects of sotatercept (MK-7962, formerly called ACE-011) treatment (plus background pulmonary arterial hypertension (PAH) therapy) versus placebo (plus background PAH therapy) on time to clinical worsening (TTCW) in participants who are newly diagnosed with PAH and are at intermediate or high risk of disease progression.

DETAILED DESCRIPTION:
This is a phase 3, randomized, double-blind, placebo-controlled study to evaluate sotatercept when added to background PAH therapy in newly diagnosed intermediate- or high risk PAH participants.

Participants enrolled in the study will have a diagnosis within 12 months of study screening of symptomatic PAH (World Health Organization (WHO) Group 1, classified as functional class (FC) II or III) and presentation of idiopathic or heritable PAH, PAH associated with connective tissue diseases (CTD), drug- or toxin- induced PAH, post shunt correction PAH, or PAH presenting at least 1 year following the correction of congenital heart defects.

As of Amendment 11, this study will be closed so that all eligible participants can receive sotatercept either on the MK-7962-004 extension study (SOTERIA, NCT04796337,) or by commercial access, if available. All eligible participants will complete the end of treatment visit before enrollment in the extension study or initiation of commercial product. Participants not enrolling into the extension study or initiating commercial product will complete the end of study visit.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants must meet all of the following criteria to be enrolled in the study:

1. Age ≥ 18 years
2. Documented diagnostic right heart catheterization (RHC) within 12 months of screening documenting a minimum PVR of ≥ 4 Wood units and pulmonary capillary wedge pressure (PCWP) or left ventricular end-diastolic pressure (LVEDP) of ≤ 15 mmHg, with the diagnosis of WHO PAH Group 1 in any of the following subtypes:

   * Idiopathic PAH
   * Heritable PAH
   * Drug/toxin-induced PAH
   * PAH associated with connective tissue disease
   * PAH associated with simple, congenital systemic to pulmonary shunts at least 1 year following repair
3. Symptomatic PAH classified as WHO FC II or III
4. Either Registry to Evaluate Early and Long-term PAH Disease Management (REVEAL) Lite 2 Risk Score ≥ 6 or Comparative, Prospective Registry of Newly Initiated Therapies for Pulmonary Hypertension (COMPERA) 2.0 risk score ≥2 (intermediate to-low-risk or above)
5. Diagnosis of PAH within 12 months of screening and on stable doses of a double or triple combination of background PAH therapies and diuretics (if any) for at least 90 days prior to screening
6. Six-minute walk distance ≥ 150 m repeated twice at screening at least 4 hours apart, but no longer than 1 week apart, and both values are within 15% of each other (calculated from the highest value)
7. Females of childbearing potential must meet the following criteria:

   * Have 2 negative urine or serum pregnancy tests as verified by the investigator prior to starting study drug administration; she must agree to ongoing urine or serum pregnancy testing during the course of the study and until 8 weeks after the last dose of the study drug
   * If sexually active with a male partner, have used highly effective contraception without interruption, for at least 28 days prior to starting the investigational product AND agreed to use the same highly effective contraception in combination with a barrier method during the study (including dose interruptions) and for 16 weeks (112 days) after discontinuation of study treatment
   * Refrain from breastfeeding a child or donating blood, eggs, or ovum for the duration of the study and for at least 16 weeks (112 days) after the last dose of study treatment
8. Male participants must meet the following criteria:

   * Agree to use a condom, defined as a male latex condom or nonlatex condom NOT made out of natural (animal) membrane (e.g., polyurethane), during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, and for at least 16 weeks (112 days) following investigational product discontinuation, even if he has undergone a successful vasectomy
   * Refrain from donating blood or sperm for the duration of the study and for 16 weeks (112 days) after the last dose of study treatment
9. Ability to adhere to study visit schedule and understand and comply with all protocol requirements
10. Ability to understand and provide written informed consent

Exclusion Criteria:

Participants will be excluded from the study if any of the following criteria are met:

1. Diagnosis of pulmonary hypertension (PH) WHO Groups 2, 3, 4, or 5
2. Diagnosis of the following PAH Group 1 subtypes: human immunodeficiency virus (HIV)-associated PAH and PAH associated with portal hypertension, schistosomiasis-associated PAH, pulmonary veno occlusive disease, and pulmonary capillary hemangiomatosis
3. Hemoglobin at screening above gender-specific upper limit of normal (ULN), per local laboratory test
4. Uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure (BP) > 180 mmHg or sitting diastolic BP > 110 mmHg during the Screening Visit after a period of rest
5. Baseline systolic BP < 90 mmHg at screening
6. Pregnant or breastfeeding women
7. Any of the following clinical laboratory values at the Screening Visit:

   * Estimated glomerular filtration rate < 30 mL/min/1.73 m2 (as defined by MDRD equation)
   * Serum alanine aminotransferase, aspartate aminotransferase, and total bilirubin levels > 3 × ULN
   * Platelet count < 50,000/mm3 (< 50.0 × 109 /L)
8. Currently enrolled in or have completed any other investigational product study within 30 days for small molecule drugs or within 5 half-lives for investigational biologics prior to the date of documented informed consent
9. Known allergic reaction to sotatercept (ACE-011), its excipients, or luspatercept
10. History of pneumonectomy
11. Pulmonary function test values of forced vital capacity < 60% predicted within 1 year prior to the Screening Visit
12. Stopped receiving any PH chronic general supportive therapy (e.g., diuretics, oxygen, anticoagulants, and digoxin) within 60 days prior to the Screening Visit
13. Initiation of an exercise program for cardiopulmonary rehabilitation within 90 days prior to the Screening Visit or planned initiation during the study (participants who are stable in the maintenance phase of a program and who will continue for the duration of the study are eligible)
14. Untreated more than mild obstructive sleep apnea
15. History of known pericardial constriction
16. History of restrictive or congestive cardiomyopathy
17. History of atrial septostomy within 180 days prior to the Screening Visit
18. Electrocardiogram with Fridericia's corrected QT interval > 500 ms during the Screening Period
19. Personal or family history of long QT syndrome or sudden cardiac death
20. Left ventricular ejection fraction < 50% on historical echocardiogram (ECHO) within 1 year prior to the Screening Visit
21. Any current or prior history of symptomatic coronary disease (prior myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft surgery, or cardiac anginal chest pain) in the past 6 months prior to the Screening Visit
22. Cerebrovascular accident within 3 months prior to the Screening Visit
23. Acutely decompensated heart failure within 30 days prior to the Screening Visit, as per investigator assessment
24. Significant (≥ 2+ regurgitation) mitral regurgitation or aortic regurgitation valvular disease
25. Received intravenous inotropes (e.g., dobutamine, dopamine, norepinephrine, and vasopressin) within 30 days prior to the Screening Visit
26. Has an active malignancy with the exception of fully excised or treated basal cell carcinoma, cervical carcinoma in-situ, or prostate cancer that is not currently or expected, during the study, to be treated with radiation therapy, chemotherapy, and/or surgical intervention, or hormonal treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Time to Clinical Worsening | Up to ~36 months
  Time to clinical worsening is defined as time from randomization to the first confirmed morbidity event or death. Clinical worsening events are defined as all-cause death, non-planned PAH-related hospitalization of ≥ 24 hours in duration, atrial septostomy, lung transplant and deterioration in performance in 6-minute walk test from baseline combined with one of the following conditions: worsening of WHO functional class from baseline, signs/symptoms of increased right heart failure, addition of a background PAH therapy or change in the background PAH therapy delivery route to parenteral. All events will be adjudicated by a blinded, independent committee of clinical experts.

SECONDARY OUTCOMES:
Percentage of Participants Achieving the Multicomponent Improvement Endpoint of 6-Minute Walk Distance (6MWD), N-terminal prohormone Btype natriuretic peptide (NT-ProBNP) and World Health Organization (WHO) Functional Class (FC) | Baseline and Week 24
  Multicomponent improvement endpoint measured by the percentage of participants achieving all of the following at Week 24 relative to baseline:
  * Improvement in 6MWD
  * Improvement or maintenance/achievement of NT-proBNP
  * Improvement in WHO FC or maintenance of WHO FC II
Percentage of Participants who Achieved a Low Registry to Evaluate Early and Long Term PAH Disease Management (REVEAL) Lite 2 Risk Score | Baseline and Week 24
  The REVEAL Lite 2 uses renal insufficiency (by estimated glomerular filtration rate (eGFR)), WHO FC, systolic blood pressure (SBP) and heart rate, 6MWD, and NT-proBNP to determine the total risk score. The scores (range: 1-14) can be defined as: low risk as a score of ≤5, intermediate risk as a score of 6 or 7, and high risk as a score of ≥8 for the survival rates.
Percentage of Participants who Maintain or Achieve a Low Simplified French Risk Score | Baseline and Week 24
  The simplified French Risk Score uses WHO FC, 6MWD, and NT-proBNP to determine the total risk score. A low risk score can be defined as attaining or maintaining all three low-risk criteria: WHO FC I or II, 6MWD > 440m, and NT-proBNP < 300 ng/L. The percentage of participants who maintain or achieve a low risk score at Week 24 versus baseline using the simplified French Risk score calculator will be reported.
Change from Baseline in NT-proBNP Levels | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to measure NT-proBNP blood concentration.
Percentage of Participants who Improve in WHO FC or Maintain WHO FC II at 24 Weeks from Baseline | Baseline and Week 24
  The severity of an individual's PAH symptoms was graded using the WHO FC system. WHO functional classification for PAH range from Class I (no limitation in physical activity, no dyspnea with normal activity), Class II (slight limitation of physical activity), Class III (marked limitation of physical activity) and Class IV (cannot perform a physical activity without any symptoms, dyspnea at rest). The change from baseline in WHO FC is classified into "Improved", "No change" and "Worsened". Improvement = reduction in FC, worsened = increase in FC and no change = no change in FC.
Change from Baseline in 6MWD | Baseline and Week 24
  The 6MWD tests the distance walked in 6 minutes as a measure of functional capacity. Change from baseline in 6MWD at Week 24 will be reported.
Overall Survival (OS) | Up to ~36 Months
  Overall survival is defined as the time from randomization to date of death due to any cause.
Change from Baseline in the Physical Impacts Domain Score of Pulmonary Arterial Hypertension Symptoms and Impact (PAH-SYMPACT)® | Baseline and Week 24
  PAH SYMPACT is a self-rating questionnaire to assess symptoms and their physical and cognitive/emotional impact. The PAH-SYMPACT® questionnaire consists of consists of 16 symptom and 25 impact items. A higher score indicates worse symptoms. Change from baseline in responses in PAH-SYMPACT questionnaire at Week 24 will be reported.
Change from Baseline in the Cardiopulmonary Symptoms Domain Score of PAH-SYMPACT® | Baseline and Week 24
  PAH SYMPACT is a self-rating questionnaire to assess symptoms and their physical and cognitive/emotional impact. The PAH-SYMPACT® questionnaire consists of consists of 16 symptom and 25 impact items. A higher score indicates worse symptoms. Change from baseline in responses in PAH-SYMPACT questionnaire at Week 24 will be reported.
Change from Baseline in the Cognitive/Emotional Impacts Domain Score of PAH-SYMPACT® | Baseline and Week 24
  PAH SYMPACT is a self-rating questionnaire to assess symptoms and their physical and cognitive/emotional impact. The PAH-SYMPACT® questionnaire consists of consists of 16 symptom and 25 impact items. A higher score indicates worse symptoms. Change from baseline in responses in PAH-SYMPACT questionnaire at Week 24 will be reported
Number of Participants who Experience an Adverse Event (AE) | Up to ~36 Months
  An AE is any untoward medical occurrence in a clinical investigation participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The number of participants who experienced an AE are presented.
Number of Participants who Discontinued Study Treatment due to AEs | Up to ~34 months
  An AE is any untoward medical occurrence in a clinical investigation participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The number of participants who discontinued study treatment due to an AE are presented.
Incidence of Anti-drug Antibodies (ADAs) to Sotatercept | Up to ~36 Months
  Blood samples collected at designated timepoints will be used to determine the ADA response to Sotatercept. The incidence of ADAs to Sotatercept over time will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (152):
- United States (28):
  - Arizona Pulmonary Specialists ( Site 1010), Scottsdale, Arizona
  - University of Arizona ( Site 1006), Tucson, Arizona
  - University of California San Diego ( Site 1002), La Jolla, California
  - UCLA Medical Center ( Site 1068), Los Angeles, California
  - University of California Irvine ( Site 1086), Orange, California
  - Santa Barbara Pulmonary Associates ( Site 1060), Santa Barbara, California
  - University of California Davis Medical Center ( Site 1064), Sherman Oaks, California
  - University of Colorado Hospital ( Site 1013), Aurora, Colorado
  - AdventHealth Medical Group Advanced Lung Disease ( Site 1058), Orlando, Florida
  - University of Iowa Hospital and Clinics ( Site 1050), Iowa City, Iowa
  - Johns Hopkins Hospital ( Site 1036), Baltimore, Maryland
  - Tufts Medical Center - PPDS ( Site 1014), Boston, Massachusetts
  - Boston Medical Center ( Site 1012), Boston, Massachusetts
  - University of Michigan ( Site 1011), Ann Arbor, Michigan
  - University of Kansas Medical Center ( Site 1020), Kansas City, Missouri
  - Washington University School of Medicine ( Site 1022), St Louis, Missouri
  - University of New Mexico, Health Sciences Center ( Site 1048), Albuquerque, New Mexico
  - NYU Langone Health ( Site 1052), New York, New York
  - University of North Carolina at Chapel Hill ( Site 1042), Chapel Hill, North Carolina
  - The Carl and Edyth Lindner Center for Research and Education at the Christ Hospital ( Site 1001), Cincinnati, Ohio
  - University of Cincinnati ( Site 1035), Cincinnati, Ohio
  - The Cleveland Clinic Foundation Taussig Cancer Center ( Site 1065), Cleveland, Ohio
  - Nazih Zuhdi Transplantation Institute ( Site 1084), Oklahoma City, Oklahoma
  - Oregon Health & Science University ( Site 1054), Portland, Oregon
  - Medical University of South Carolina ( Site 1003), Charleston, South Carolina
  - Vanderbilt University Medical Center ( Site 1027), Nashville, Tennessee
  - University of Texas Southwestern Medical Center ( Site 1038), Dallas, Texas
  - University of Utah ( Site 1049), Salt Lake City, Utah
- Argentina (12):
  - Cardiologia Palermo ( Site 1911), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro Medico Dra De Salvo ( Site 1904), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral ( Site 1901), Pilar, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes ( Site 1903), Quilmes, Buenos Aires
  - Instituto De Enfermedades Respiratorias E Investigacion Medica ( Site 1910), Villa Vatteone, Buenos Aires
  - Instituto Médico DAMIC ( Site 1909), Córdoba, Córdoba Province
  - Instituto Medico Rio Cuarto ( Site 1907), Río Cuarto, Córdoba Province
  - Hospital Provincial del Centenario ( Site 1912), Rosario, Santa Fe Province
  - Instituto Cardiovascular de Rosario ( Site 1906), Rosario, Santa Fe Province
  - Sanatorio Parque ( Site 1905), Rosario, Santa Fe Province
  - Sanatorio Allende ( Site 1908), Córdoba
  - Hospital Provincial Dr. Jose M. Cullen ( Site 1902), Santa Fe
- Australia (7):
  - Royal Prince Alfred Hospital ( Site 1106), Camperdown, New South Wales
  - John Hunter Hospital ( Site 1101), Newcastle, New South Wales
  - Prince Charles Hospital ( Site 1104), Chermside, Queensland
  - Princess Alexandra Hospital ( Site 1108), Woolloongabba, Queensland
  - Royal Adelaide Hospital ( Site 1109), Adelaide, South Australia
  - Royal Hobart Hospital ( Site 1107), Hobart, Tasmania
  - Fiona Stanley Hospital ( Site 1103), Murdoch, Western Australia
- Austria (4):
  - Medizinische Universität Graz ( Site 2003), Graz, Styria
  - Medizinische Universitat Innsbruck ( Site 2004), Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Elisabethinen ( Site 2002), Linz, Upper Austria
  - Medizinische Universitat Wien ( Site 2001), Vienna, Vienna
- Belgium (2):
  - Hopital Erasme ( Site 1402), Anderlecht, Bruxelles-Capitale, Region de
  - UZ Gasthuisberg ( Site 1401), Leuven, Vlaams-Brabant
- Brazil (4):
  - Hospital Madre Teresa ( Site 1804), Belo Horizonte, Minas Gerais
  - Irmandade da Santa Casa de Misericordia de Porto Alegre ( Site 1805), Porto Alegre, Rio Grande do Sul
  - Hospital Sao Paulo ( Site 1806), São Paulo, São Paulo
  - Instituto do Coracao - HCFMUSP ( Site 1803), São Paulo
- Canada (4):
  - University of Alberta Hospital ( Site 2101), Edmonton, Alberta
  - St Boniface General Hospital ( Site 2106), Winnepeg, Manitoba
  - McMaster University - HSC ( Site 2105), Hamilton, Ontario
  - Sir Mortimer B Davis Jewish General Hospital ( Site 2103), Montreal, Quebec
- Colombia (4):
  - Centro Cardiovascular Colombiano Clínica Santa María Clínica Cardio VID ( Site 3402), Medellín, Antioquia
  - Fundacion Neumologica Colombiana ( Site 3403), Bogota, Cundinamarca
  - Fundacion Valle Del Lili ( Site 3401), Cali, Valle del Cauca Department
  - Centro Medico Imbanaco de Cali S.A ( Site 3404), Cali, Valle del Cauca Department
- Croatia (2):
  - University Hospital Centre Split city ( Site 3901), Split, Split-Dalmatia County
  - Klinicki Bolnicki Centar Zagreb ( Site 3902), Zagreb, Zagreb County
- Czechia (2):
  - Institut Klinicke a Experimentalni Mediciny ( Site 2202), Prague, Praha 4
  - Vseobecna fakultni nemocnice v Praze ( Site 2201), Prague
- Denmark (2):
  - Rigshospitalet ( Site 3802), København Ø, Capital Region
  - Aarhus Universitetshospital, Skejby ( Site 3801), Aarhus, Central Jutland
- France (15):
  - Hopital Louis Pasteur ( Site 1311), Nice, Alpes-Maritimes
  - Hopital Louis Pradel ( Site 1317), Lyon, Auvergne
  - Hopitaux Universitaires de Strasbourg ( Site 1307), Strasbourg, Bas-Rhin
  - Hopital Cavale Blanche ( Site 1314), Brest, Brittany Region
  - CHU Caen Normandie ( Site 1325), Caen, Calvados
  - CHU de Besancon ( Site 1303), Besançon, Doubs
  - Hopital Haut Leveque ( Site 1312), Bordeaux, Gironde
  - CHU de Toulouse - Hopital Larrey ( Site 1315), Toulouse, Haute-Garonne
  - C.H.U. de Tours - Hopital Bretonneau ( Site 1310), Tours, Indre-et-Loire
  - Hopital Nord Laennec ( Site 1309), Nantes, Loire-Atlantique
  - CHU Angers ( Site 1313), Angers, Maine-et-Loire
  - C.H.U. de Nancy. Hopital de Brabois Adultes ( Site 1308), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre Hospitalier Universitaire de Saint-Etienne ( Site 1302), Saint-Priest-en-Jarez, Pays de la Loire Region
  - CHU - Hopital de Bicetre ( Site 1304), Le Kremlin-Bicêtre, Val-de-Marne
  - CHU de Poitiers ( Site 1316), Poitiers, Vienne
- Germany (11):
  - Universitaetsklinikum Heidelberg ( Site 1509), Heidelberg, Baden-Wurttemberg
  - Krankenhaus Neuwittelsbach ( Site 1510), Munich, Bavaria
  - Universitaetsklinik Regensburg ( Site 1503), Regensburg, Bavaria
  - Medizinische Hochschule Hannover ( Site 1505), Hanover, Lower Saxony
  - Universitaetsklinikum Giessen und Marburg GmbH ( Site 1512), Bad Oeynhausen, North Rhine-Westphalia
  - Uniklinik Köln ( Site 1511), Cologne, North Rhine-Westphalia
  - Universitatsklinikum des Saarlandes ( Site 1513), Homburg, Saarland
  - Universitaetsklinikum Carl Gustav Carus ( Site 1501), Dresden, Saxony
  - Universitatsklinikum Leipzig ( Site 1508), Leipzig, Saxony
  - Universitaetsklinik und Poliklinik Halle/Saale ( Site 1502), Halle, Saxony-Anhalt
  - DRK Kliniken Berlin Westend ( Site 1507), Berlin
- Greece (4):
  - Evangelismos General Hospital of Athens ( Site 3605), Athens, Attica
  - Onassis Cardiac Surgery Center ( Site 3602), Athens, Attica
  - Attikon University General Hospital of Athens ( Site 3604), Haidari, Attica
  - AHEPA University General Hospital of Thessaloniki ( Site 3601), Thessaloniki
- Israel (4):
  - Assuta Ashdod Medical Center ( Site 1710), Ashdod
  - Lady Davis Carmel Medical Center ( Site 1705), Haifa
  - Hadassah Medical Center ( Site 1711), Jerusalem
  - Sheba Medical Center ( Site 1701), Tel Litwinsky
- Italy (5):
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) ( Site 2405), Trieste, Friuli Venezia Giulia
  - Ospedale S. Giuseppe Multimedica ( Site 2403), Milan, Lombardy
  - Azienda Ospedaliera San Gerardo di Monza ( Site 2406), Monza, Monza E Brianza
  - Azienda Ospedaliera R. N. V. Monaldi ( Site 2407), Napoli
  - La Sapienza-Università di Roma-Policlinico Umberto I ( Site 2402), Roma
- Netherlands (4):
  - Radboud University Nijmegen Medical Centre ( Site 2605), Nijmegen, Gelderland
  - Maastricht University Medical Center ( Site 2603), Maastricht, Limburg
  - VU Medisch Centrum ( Site 2601), Amsterdam, North Holland
  - Erasmus MC ( Site 2604), Rotterdam, South Holland
- Waikato District Health Board ( Site 2702), Hamilton, Waikato Region, New Zealand
- Poland (2):
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II ( Site 2801), Krakow, Lesser Poland Voivodeship
  - Instytut Gruzlicy i Chorob Pluc w Warszawie ( Site 2802), Warsaw, Masovian Voivodeship
- Portugal (3):
  - Hospital Garcia de Orta ( Site 3501), Almada, Setúbal District
  - Centro Hospitalar E Universitário De Coimbra ( Site 3502), Coimbra
  - Hospital Pulido Valente ( Site 3503), Lisbon
- Serbia (4):
  - Clinical Center of Serbia ( Site 2901), Belgrade, Beograd
  - Institute for pulmonary diseases of Vojvodina ( Site 2906), Kamenitz, Juznobacki Okrug
  - University Clinical Center Nis ( Site 2904), Niš, Nisavski Okrug
  - Clinical Center Kragujevac ( Site 2905), Kragujevac, Sumadijski Okrug
- South Korea (6):
  - Gachon University Gil Medical Center ( Site 3103), Namdong-Gu, Incheon
  - Chonnam National University Hospital ( Site 3105), Gwangju, Kyonggi-do
  - Samsung Medical Center ( Site 3106), Seuol, Seoul
  - Seoul National University Hospital ( Site 3102), Seoul
  - Severance Hospital Yonsei University Health System - PPDS ( Site 3101), Seoul
  - The Catholic University of Korea St. Mary s Hospital ( Site 3104), Seoul
- Spain (8):
  - Hospital Universitario de Son Espases ( Site 1611), Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marques de Valdecilla ( Site 1601), Santander, Cantabria
  - Hospital Universitario Puerta de Hierro (Majadahonda) ( Site 1604), Majadahonda, Madrid
  - Hospital Universitari Vall de Hebron ( Site 1605), Barcelona
  - Hospital Universitario 12 de Octubre ( Site 1603), Madrid
  - Hospital Universitario La Paz ( Site 1610), Madrid
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca ( Site 1608), Salamanca
  - Hospital Virgen de la Salud ( Site 1607), Toledo
- Sweden (3):
  - Skanes Universitetssjukhus Lund ( Site 3203), Lund, Skåne County
  - Hjart-lungmedicin och klinisk fysiologi ( Site 3204), Uppsala, Uppsala County
  - Norrlands Universitetssjukhus ( Site 3205), Umeå, Västerbotten County
- UniversitätsSpital Zürich ( Site 3301), Zurich, Switzerland
- Taiwan (3):
  - Kaohsiung Veterans General Hospital ( Site 3702), Kaohsiung City
  - China Medical University Hospital ( Site 3701), Taichung
  - National Cheng Kung University Hospital ( Site 3703), Tainan
- United Kingdom (7):
  - Papworth Hospital NHS Foundation Trust ( Site 1208), Cambrigge, Cambridgeshire
  - Sheffield Teaching Hospital NHS Foundation Trust ( Site 1207), Sheffield, Derbyshire
  - Golden Jubilee National Hospital ( Site 1204), Glasgow, Glasgow City
  - Royal Free London NHS Foundation Trust ( Site 1202), London, London, City of
  - Royal Brompton Hospital ( Site 1206), London, London, City of
  - Imperial College Healthcare NHS Trust ( Site 1203), London, London, City of
  - Freeman Hospital ( Site 1205), Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] McLaughlin VV, Hoeper MM, Badesch DB, Ghofrani HA, Gibbs JSR, Gomberg-Maitland M, Preston IR, Souza R, Waxman AB, Kopec G, Meyer G, Olsson KM, Fu W, Shi Y, Miller B, Kim SS, Mackenzie HS, Brambatti M, Patel MJ, Koglin J, Cornell AG, Humbert M; HYPERION Trial Investigators. Sotatercept for Pulmonary Arterial Hypertension within the First Year after Diagnosis. N Engl J Med. 2025 Oct 23;393(16):1599-1611. doi: 10.1056/NEJMoa2508170. Epub 2025 Sep 30. PMID 41025556
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26123&tenant=MT_MSD_9011